CLINICAL TRIAL: NCT06432699
Title: Rate of Canine Retraction and Pain Perception Following Micro-osteoperforation- a Split
Brief Title: Rate of Canine Retraction and Pain Perception Following Micro-osteoperforation- a Split Mouth Clinical Study
Acronym: MOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Shoaib Rahim, ZAINAB BUTT, Foundation University Islamabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FF/FUMC/215-372Phy/23
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-06

CONDITIONS: Pain; Rate of Canine Retraction
Keywords: MOP
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a single-blind, randomized parallel-arm study with two arms. Participants will be randomly assigned to either MOPS or no Mops
Masking Description: Participants will be randomly assigned to receive Micro-osteoperforation and the other side will be control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this arm will receive no MOP treatment
- Experimental (Experimental): participants in this arm will receive MOPS intervention
  Interventions: Other: micro osteoperforation

INTERVENTIONS:
Other: micro osteoperforation — one side used for mops while other side will be control in same patient
  Other Names: Placebo/Controlled
  Arms: Experimental

SUMMARY:
DEFINITION: A short description of clinical study , including a brief statement of clinical study's hypothesis, written in language intended for the lay public Limit: 5000 CHARACTERS

DETAILED DESCRIPTION:
Definition: Extended description of the protocol ,including more technical information(as compared to the brief Summary), if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures.

Limit:32,000 characters. For Patient Registries: Also describe the applicable registry procedures and other quality factors (for examples, third party certification, on site audit). In particular , summarize any procedures implemented as part of the patient registry, including , but not limited to the following:

* Quality assurance plan that addresses data validation and registry procedures, including and plans for site monitoring and auditing
* Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
* Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources( for example, medical records, paper or electronic case reports forms, or interactive voice response systems)
* Data Dictionary that contains detailed descriptions of each variable used by the registry, including, including the source of the variable, coding information if used (for example World Health Organization Drug Dictionary, MedDRA), and normal ranges if relevant.
* STANDARD OPERATING PROCEDURE TO ADDRESS REGISTRY REGISTRY OPERATIONS AND ANALYSISACTIVITIES, SUCH AS PATIENT RECRUITMENT DATA COLLECTION,DATA MANAGEMENT., DATA ANALYSIS, reporting for adverse events, and change management.
* Sample Size Assessment to specify the number of participants or participate years necessary to demonstrate an effect.
* Plan for missing data to address situations where variable are reported a missing , unavailable non-reported, interpretable, or considered missing because of data inconsistency or out-of-range results.
* Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives , as specified in the study protocol or plan

ELIGIBILITY:
Inclusion Criteria:

- 1. Age range around 15-40 years. 2. Patients which have class I malocclusion or class II Div I malocclusion and include first premolar extraction as part of treatment plan..

3. No orthodontic treatment previously 4. Radiographic evidence showing no bone loss 5. History showing no periodontal disease. 6. History showing no systemic disease. 7. Probing depth less than 4 mm across the entire dentition 8. No active carious lesion or any sign of gingivitus

Exclusion Criteria:

1. Presence of any craniofacial abnormality.
2. Any history of bleeding disorders.
3. Poor oral hygiene.
4. Use of bisphosphonates, analgesics, anti-inflammatory drugs, corticosteroids for more than three months prior to treatment or during treatment.
5. Active diseases such as metabolic bone disease.
6. Malocclusions requiring surgical intervention.
7. Smoker

   -

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
pain will be measured after intervention of visual analogue scale | three months since the MOPS
  patient after undergoing micro-osteoperforation will be aske to measure pain and check rate of canine retraction

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan

REFERENCES:
- [Background] 1. Kundi, I., Alam, M. K., & Shaheed, S. (2020). Micro-osteo perforation effects as an intervention on canine retraction. The Saudi dental journal, 32(1), 15-20. https://doi.org/10.1016/j.sdentj.2019.05.009 2. Husain S, Sundari S. Comparison of the effectiveness of piezocision-aided canine retraction augmented with micro-osteoperforation: a randomized controlled trial. Angle Orthod. 2023 Oct 16. doi: 10.2319/052323-370.1. Epub ahead of print. PMID: 37839802. 12 3. Aboalnaga AA, Aboalnaga AA, Salah Fayed MM, El-Ashmawi NA, Soliman SA. Effect of micro-osteoperforation on the rate of canine retraction: a split- mouth randomized controlled trial. Prog Orthod. 2019 Jun;20(1) 21. doi:10.1186/s40510-019-0274-0. PMID: 31155698; PMCID: PMC6545296. 4. Bolat Gümüş, E., Kınsız, E. Effects of miniscrew-facilitated micro- osteoperforations on the rate of orthodontic tooth movement. J Orofac Orthop 84 (Suppl 2), 104-110 (2023). 5. Martina K., Kumar P., Misra V., Attri S., Yadav A., Sam R., Kumar R.. To evaluate the rate of canine retraction and pain perception following micro- osteoperforation - a split-mouth clinical study. Australasian Orthodontic Journal. 2022;38(2): 388-395